CLINICAL TRIAL: NCT01301833
Title: Long-term Safety Study of MP-513 as Monotherapy or in Combination With Oral Antihyperglycaemic Agent in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: Long-term Safety Study of MP-513 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3000-A14
Record Dates: First submitted 2011-02-14; First posted 2011-02-23 (Estimated); Results first posted 2015-08-28 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine; Biguanides; Glycoside Hydrolase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- teneligliptin (Experimental): teneligliptin (20 mg once daily, titrated to 40 mg if no adequate efficacy is obtained )
  Interventions: Drug: teneligliptin
- teneligliptin and glinide (Experimental): teneligliptin (20 mg once daily, titrated to 40 mg if no adequate efficacy is obtained ) plus glinide
  Interventions: Drug: teneligliptin; Drug: glinide
- teneligliptin and biguanide (Experimental): teneligliptin (20 mg once daily, titrated to 40 mg if no adequate efficacy is obtained ) plus biguanide
  Interventions: Drug: teneligliptin; Drug: biguanide
- teneligliptin and alpha-glucosidase inhibitor (Experimental): teneligliptin (20 mg once daily, titrated to 40 mg if no adequate efficacy is obtained ) plus alpha-glucosidase inhibitor
  Interventions: Drug: teneligliptin; Drug: alpha-glucosidase inhibitor

INTERVENTIONS:
Drug: teneligliptin
  Other Names: MP-513
Drug: glinide
  Arms: teneligliptin and glinide
Drug: biguanide
  Arms: teneligliptin and biguanide
Drug: alpha-glucosidase inhibitor
  Arms: teneligliptin and alpha-glucosidase inhibitor

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of MP-513 (Teneligliptin) as monotherapy or in combination with oral antihyperglycaemic agent in patients with type 2 Diabetes for 52 weeks administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients who has been receiving a stable dose and regimen of oral antihyperglycaemic agent (biguanide agent,α-glucosidase inhibitor,rapid insulin secretagogue) for diabetes over 12 weeks before administration of investigational drug
* Patients who are under dietary management and taking therapeutic exercise for diabetes over 12 weeks before administration of investigational drug
* Patients whose HbA1c is between 6.5% - 10.0%
* Patients who were not administered diabetes therapeutic drugs prohibited for concomitant use within 12 weeks before administration of investigational drug

Exclusion Criteria:

* Patients with type 1 diabetes, diabetes mellitus caused by pancreas impairment, or secondary diabetes (Cushing disease, acromegaly, etc)
* Patients who are accepting treatments of arrhythmias
* Patients with serious diabetic complications
* Patients who are habitual excessive alcohol consumption.
* Patients with severe hepatic disorder or severe renal disorder.
* Patients who are pregnant, lactating, and probably pregnant patients, and patients who can not agree to contraception

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Kadowaki, Professor, Study Director — Tokyo University; Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (1):
- Chitose-shi, Hokkaido, Japan

REFERENCES:
- [Result] Kadowaki T, Marubayashi F, Yokota S, Katoh M, Iijima H. Safety and efficacy of teneligliptin in Japanese patients with type 2 diabetes mellitus: a pooled analysis of two Phase III clinical studies. Expert Opin Pharmacother. 2015 May;16(7):971-81. doi: 10.1517/14656566.2015.1032249. Epub 2015 Apr 10. PMID 25861982

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Teneligliptin | Teneligliptin and Glinide | Teneligliptin and Biguanide | Teneligliptin and Alpha-glucosidase Inhibitor
Started | 212 | 80 | 95 | 75
Completed | 197 | 72 | 88 | 68
Not Completed | 15 | 8 | 7 | 7
Not completed — Adverse Event | 7 | 5 | 5 | 5
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Not completed — Physician Decision | 3 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 2
Not completed — Personal matter | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teneligliptin | Teneligliptin and Glinide | Teneligliptin and Biguanide | Teneligliptin and Alpha-glucosidase Inhibitor | Total
Number analyzed (Participants) | 212 | 80 | 95 | 75 | 462
Age, Customized [Number; unit: participants]
  <65 years | 141 | 45 | 66 | 39 | 291
  >=65 years | 71 | 35 | 29 | 36 | 171
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 31 | 37 | 25 | 164
  Male | 141 | 49 | 58 | 50 | 298

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Treatment-emergent adverse events (TEAE) were defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through 14 days after receiving the last dose of study drug.
Time Frame: 52 Weeks
Population: Safety set, consisting of all patients, who received at least one dose of study drug and who had at least one safety data after the treatment of study drug.
Measure: Number; unit: participants
Arm/Group | Teneligliptin | Teneligliptin and Glinide | Teneligliptin and Biguanide | Teneligliptin and Alpha-glucosidase Inhibitor
Number analyzed (Participants) | 212 | 80 | 95 | 75
participants
  Serious Adverse Event | 14 | 3 | 6 | 6
  Other Adverse Event | 182 | 72 | 81 | 59

2. Secondary Outcome: Change From Baseline in HbA1c at Week 52
Time Frame: Baseline and 52 weeks
Population: The full analysis set, consisting of all type 2 diabetic patients, who received at least one dose of study drug and who had at least one efficacy data after the treatment of study drug. Analysis based on last observation carried forward, where the last postbaseline observed value was carried forward and used for Week 52 where data was missing.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Teneligliptin | Teneligliptin and Glinide | Teneligliptin and Biguanide | Teneligliptin and Alpha-glucosidase Inhibitor
Number analyzed (Participants) | 212 | 80 | 95 | 75
Percent | -0.63 (0.64) | -0.76 (0.70) | -0.78 (0.75) | -0.89 (0.64)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 52
Time Frame: Baseline and 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg / dL
Arm/Group | Teneligliptin | Teneligliptin and Glinide | Teneligliptin and Biguanide | Teneligliptin and Alpha-glucosidase Inhibitor
Number analyzed (Participants) | 212 | 80 | 95 | 75
mg / dL | -11.7 (25.5) | -13.7 (23.7) | -12.7 (27.1) | -19.5 (23.5)

4. Secondary Outcome: Change From Baseline in Fasting Glucagon at Week 52
Time Frame: Baseline and 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg / mL
Arm/Group | Teneligliptin | Teneligliptin and Glinide | Teneligliptin and Biguanide | Teneligliptin and Alpha-glucosidase Inhibitor
Number analyzed (Participants) | 212 | 80 | 95 | 75
pg / mL | 2.8 (12.5) | 5.3 (13.7) | 5.0 (14.4) | 6.9 (15.2)

5. Secondary Outcome: Change From Baseline in Fasting Immuno Reactive Insulin (IRI) at Week 52
Time Frame: Baseline and 52 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μU / mL
Arm/Group | Teneligliptin | Teneligliptin and Glinide | Teneligliptin and Biguanide | Teneligliptin and Alpha-glucosidase Inhibitor
Number analyzed (Participants) | 212 | 80 | 95 | 75
μU / mL | 0.988 (8.314) | 0.211 (2.378) | -0.173 (9.093) | -0.330 (2.713)

ADVERSE EVENTS:
Arm/Group | Teneligliptin | Teneligliptin and Glinide | Teneligliptin and Biguanide | Teneligliptin and Alpha-glucosidase Inhibitor
Serious Adverse Events (participants affected / at risk) | 14/212 | 3/80 | 6/95 | 6/75
Other Adverse Events (participants affected / at risk) | 182/212 | 72/80 | 81/95 | 59/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teneligliptin (N=212) | Teneligliptin and Glinide (N=80) | Teneligliptin and Biguanide (N=95) | Teneligliptin and Alpha-glucosidase Inhibitor (N=75)
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ota's naevus (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Thyroiditis (Endocrine disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 2 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teneligliptin (N=212) | Teneligliptin and Glinide (N=80) | Teneligliptin and Biguanide (N=95) | Teneligliptin and Alpha-glucosidase Inhibitor (N=75)
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 1 | 1 | 1 | 0
Body tinea (Infections and infestations) | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 7 | 7 | 5 | 2
Cellulitis orbital (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 6 | 1 | 5 | 2
Dermatitis infected (Infections and infestations) | 0 | 2 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 3 | 2 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 3 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 3 | 0 | 0 | 0
Influenza (Infections and infestations) | 3 | 4 | 3 | 2
Mumps (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 62 | 19 | 28 | 21
Onychomycosis (Infections and infestations) | 4 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 12 | 4 | 5 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 1 | 1 | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 4 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 2 | 0
Urethritis (Infections and infestations) | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Vulvitis (Infections and infestations) | 0 | 1 | 0 | 0
Peritonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Gingival abscess (Infections and infestations) | 1 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 | 1 | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 1 | 0 | 1
Mycoplasma infection (Infections and infestations) | 0 | 0 | 0 | 1
Dental gangrene (Infections and infestations) | 1 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 3 | 0 | 0 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 2 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 4 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Dysphoria (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 2 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 2 | 1 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 3 | 0 | 1
Headache (Nervous system disorders) | 5 | 0 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 1 | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 1 | 1 | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0 | 0 | 0
Asthenopia (Eye disorders) | 4 | 0 | 0 | 0
Astigmatism (Eye disorders) | 1 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 6 | 2 | 2 | 0
Chalazion (Eye disorders) | 0 | 0 | 2 | 0
Conjunctival cyst (Eye disorders) | 0 | 0 | 1 | 0
Conjunctival deposit (Eye disorders) | 1 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 4 | 0 | 0 | 2
Diabetic retinopathy (Eye disorders) | 1 | 1 | 2 | 1
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 2 | 0 | 0 | 0
Iritis (Eye disorders) | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 2 | 0 | 1 | 0
Open angle glaucoma (Eye disorders) | 2 | 0 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Retinal tear (Eye disorders) | 2 | 0 | 0 | 1
Pingueculitis (Eye disorders) | 1 | 0 | 0 | 0
Conjunctivochalasis (Eye disorders) | 0 | 0 | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0 | 0
Normal tension glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 1 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 3 | 1 | 0 | 0
Peripheral coldness (Vascular disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 20 | 11 | 10 | 8
Allergic pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 2 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 3 | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 7 | 2 | 7 | 2
Dental caries (Gastrointestinal disorders) | 2 | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 0 | 2 | 4
Duodenal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 2 | 3 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 3 | 2 | 4 | 3
Gastritis atrophic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3 | 4 | 5
Gingivitis (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 5 | 1 | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Periodontal disease (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Periodontitis (Gastrointestinal disorders) | 7 | 3 | 3 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 3 | 1
Tooth loss (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 2 | 0
Hepatic steatosis (Hepatobiliary disorders) | 2 | 2 | 3 | 1
Gallbladder polyp (Hepatobiliary disorders) | 2 | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 | 0 | 3 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 8 | 4 | 1 | 7
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 2 | 4 | 4
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 2 | 3 | 2
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 3
Periarthritis (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3 | 2
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 2 | 2 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 2 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1
IgA nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 3 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 3 | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0 | 2 | 3
Amylase increased (Investigations) | 2 | 2 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 2 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 12 | 4 | 6 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 1 | 0
Blood potassium increased (Investigations) | 2 | 2 | 0 | 1
Blood pressure increased (Investigations) | 2 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 2 | 1 | 2 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 3 | 0 | 2 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | 2 | 1
Glucose urine present (Investigations) | 10 | 3 | 7 | 0
Blood urine present (Investigations) | 15 | 6 | 9 | 5
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 3 | 1 | 4 | 2
Low density lipoprotein increased (Investigations) | 0 | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 0 | 1
Protein urine present (Investigations) | 14 | 6 | 4 | 5
Urine ketone body present (Investigations) | 7 | 6 | 6 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 2
Occult blood positive (Investigations) | 0 | 1 | 1 | 0
Helicobacter test positive (Investigations) | 0 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 3 | 3 | 2 | 0
Bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Chillblains (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 2
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 10 | 5 | 4 | 3
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Open wound (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 4
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0
Heat illness (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other